CLINICAL TRIAL: NCT01700881
Title: A Nutrition Intervention for Arthritis-2
Brief Title: A Nutrition Intervention for Arthritis -2
Acronym: WCCR-ARTH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WCCR-ARTH-2
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Diet, Fat-Restricted, Diet, Vegetarian
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Diet, Plant-Based; Diet, Vegan; Dietary Supplements; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plant-based diet (Experimental): The diet group will be asked to follow a low-fat, vegan diet for 16 weeks
  Interventions: Other: Plant-based diet
- Supplement (Placebo Comparator): The supplement group will follow an unrestricted diet, but will be given a pill containing a small, clinically insignificant amount of omega- 3 oils and vitamin E, which will serve as a placebo.
  Interventions: Other: Supplement

INTERVENTIONS:
Other: Plant-based diet — Weekly instructions will be given to the participants in the intervention group about following vegan diet.
  Other Names: Vegan diet
  Arms: Plant-based diet
Other: Supplement — Unrestricted diet with clinically insignificant amount of omega- 3 oils and vitamin E
  Other Names: Vitamin E
  Arms: Supplement

SUMMARY:
The purpose of the study is to assess whether, in individuals with rheumatoid arthritis, a low-fat, vegan diet improves pain and other subjective symptoms more effectively than a control supplement or a placebo. The principal measure is pain as measured by Visual Analog Scale (VAS) and disease activity as measured by number of painful swollen and tender joints, respectively. The study duration is 36 weeks.

This study tests that a low fat, plant-based (vegan) diet free of foods commonly identified as triggers improves mood, using the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R), and the Beck Depression Inventory II (BDI-II).

DETAILED DESCRIPTION:
Preliminary evidence suggests that low-fat, vegetarian diets and certain nutritional supplements can help reduce pain and also reduce the need for pain medications for some people. The investigators will ask about 100 people to participate. All of them will get a low-fat, vegan diet and a nutritional supplement (mixture of omega-3 oils and vitamin E or a placebo), although some will get the diet first, and others will get the supplement first. This order in which they will get the diet and the supplement will be determined randomly, that is, by chance (like the toss of a coin). The principal measure is pain as measured by Visual Analog Scale (VAS) and disease activity as measured by number of painful swollen and tender joints, respectively. The Beck Depression Inventory II (BDI-II)will be used to measure changes in mood. The study duration is 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of rheumatoid arthritis based on 2010 ACR / EULAR Rheumatoid Arthritis Classification Criteria. Classification as "definite RA" is based on:

* the confirmed presence of synovitis in at least 1 joint
* absence of an alternative diagnosis that better explains the synovitis
* and achievement of a total score of 6 or greater (of a possible 10): 24 Joint involvement, designating the metacarpophalangeal joints, proximal interphalangeal joints, the interphalangeal joint of the thumb, second through third metatarsophalangeal joint and wrist as small joints, and elbows, hip joints and knees as large joints:

  1. Involvement of 1 large joint gives 0 points
  2. Involvement of 2-10 large joints gives 1 point
  3. Involvement of 1-3 small joints (with or without involvement of large joints) gives 2 points
  4. Involvement of 4-10 small joints (with or without involvement of large joints) gives 3 points
  5. Involvement of more than 10 joints (with involvement of at least 1 small joint) gives 5 points
* Serological parameters - including the rheumatoid factor as well as anti-citrullinated protein antibody (ACPA):

  1. Negative RF and negative ACPA gives 0 points
  2. Low-positive RF or low-positive ACPA gives 2 points
  3. High-positive RF or high-positive ACPA gives 3 points Acute phase reactants: 1 point for elevated erythrocyte sedimentation rate (ESR) or elevated C-reactive protein (CRP) value Duration of arthritis: 1 point for symptoms lasting six weeks or longer
* Continuing or recurring pain (i.e., joint pain daily, unless on pain medication).
* Age at least 18 years
* Ability and willingness to participate in all components of the study
* Willingness to be assigned to either the diet group or supplement group
* Pain medications unchanged within last 6 weeks.

Exclusion Criteria:

* < 18 years of age
* Rheumatoid arthritis for more than 6 years
* Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
* Use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
* Pregnancy
* Unstable medical or psychiatric illness
* Likely to be disruptive in group sessions (as determined by research staff)
* Already following a low-fat, vegan diet
* Lack of English fluency
* Inability to maintain current medication regimen
* Inability or unwillingness to participate in all components of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10-01; Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Pain Score | Change in pain score from Baseline at 4 months
  will be measured by visual analog scale
Disease Activity score | Change in disease activity score from Baseline at 4 months
  measured by number of painful, swollen and tender joints
Improvement in mood | Change in mood from Baseline at 4 months
  measured by the Beck Depression Inventory II (BDI-II).
Improvement in depression | Change in depression from Baseline at 4 months
  measured by Epidemiologic Studies Depression Scale-Revised (CESD-R).

SECONDARY OUTCOMES:
Quality of Life regarding pain | Change in quality of life from Baseline at 4 months
  Measured by a modified health assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Barnard ND, Levin S, Crosby L, Flores R, Holubkov R, Kahleova H. A Randomized, Crossover Trial of a Nutritional Intervention for Rheumatoid Arthritis. Am J Lifestyle Med. 2022 Apr 3;19(2):266-275. doi: 10.1177/15598276221081819. eCollection 2025 Feb. PMID 39981557